CLINICAL TRIAL: NCT07186257
Title: Impact of Uterine Leiomyoma Location on Uterine Artery Doppler Velocimetry : a Prospective Cohort Study
Brief Title: Impact of Uterine Leiomyoma Location on Uterine Artery Doppler Velocimetry
Acronym: ULLADS
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, İlke Esin Aydıner, Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2024-11-17
Record Dates: First submitted 2025-06-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Leiomyoma (Uterine Fibroids)
Keywords: leiomyoma; uterine artery; doppler ultrasound; doppler velocimetry; uterine leiomyoma; leiomyoma location
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- submucous leiomyoma: patients who are diagnosed with submucous leiomyoma
- intramural leiomyoma: patients who are diagnosed with intramural leiomyoma
- subserous leiomyoma: patients who are diagnosed with subserous leiomyoma
- control: patients in the control group

SUMMARY:
Aim: Investigation of the impact of uterine leiomyoma location on uterine artery velocimetry Materials and Methods: It is a single-center prospective cohort study. The information regarding patients' demography, medical history, obstetric history, menstrual patterns, gynecological history, patients' complaints and physical examination recorded. For the patients who experience pain, visual analog scores were recorded. Total number of 185 patients have been administered for this study. They are further divided into four sub-groups according to the leiomyoma location. All measurements were recorded by the same doppler ultrasonography machine and same preset settings were used for each measurement. All examinations were performed by the same investigator. The measurements of uterus and myoma in ortogonal projections were recorded to calculate the volume by the prolate elipsoid formula. The location of each myoma were noted according to the FIGO classification. The recorded doppler ultrasonography indices included pulsatility index, resistance index and sistol/diastol ratio. IBM SPSS 27.0.0 was used for statistical analysis.

Results: Mean values of PI, RI and S/D ratio were significantly lower in intramural myoma subgroup (p<0,01). The doppler parameters were significantly higher for submucousal myoma compared to intramural and subserous myoma groups (p<0,01) while there was no significant difference with control group. The impact of uterin leiomyoma location on uterin arter doppler findings were not altered by the effects of demographical features, age, BMI or history of c-section. The increased volumes of both uterus and myoma negatively correlated with the doppler indices while the history of c-section had a positive correlation with the doppler findings. The complaints of the patients at admission showed no effect on the doppler parameters.

Conclusion: The uterin leiomyoma location has been showed to be significant factor on uterin doppler velocimetry. The leiomyomas with intramural component significantly decreased the resistance in uterine artery. Further research is required to fully understand the underlying mechanism.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years old
* accepting the transvaginal ultrasound examination and having no impediment of having transvaginal ultrasound examination
* premenopausal status
* giving verbal and written consent to enroll
* being in the follicular phase of the menstrual cycle

Exclusion Criteria:

* being younger than 18 years old
* pregnancy or postpartum status
* postmenopausal status
* being virgin
* not accepting the transvaginal ultrasound examination or having an impeding condition
* having a disease causing circulaiton abnormalities, cardiac diseases, or other comorbidities effecting circulation
* diagnosed diabetes
* taking any of the hormonal drugs (such as oral contraceptives, levonorgestrel realisng intrauterine devices)
* diagnosed with any other gyneoclogical pathologies ( adenomyosis, endometriosis, adnexial masses, gynecologic malignancies, pelvic inflammatory diseases etc. )
* being in the phases of menstrual cycle other than follicular phase
* diagnosis with type 2-5 and type 8 leiomyoma uteri according to the FIGO classification
* having multiple uterine leiomyomas
* having a uterine leiomyoma larger than 500cm3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients who have appointments for the outpatient clinic of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
the impact of uterine leiomyom location on uterine artery pulsatility index (PI) | The doppler measurement is performed at the enrollment of the first patient up to one year
  The pulsatility index (PI) measurements compared amongst the study groups of different leiomyoma localizations (submucous, intramural, subserous) and control group
the impact of uterine leiomyom location on uterine artery resistance index (RI) | The doppler measurement is performed at the enrollment of the first patient up to one year
  The resistance index (RI) measurements compared amongst the study groups of different leiomyoma localizations (submucous, intramural, subserous) and control group
the impact of uterine leiomyom location on uterine artery systolic/diastolic ratio (S/D) | The doppler measurement is performed at the enrollment of the first patient up to one year
  The systolic/diastolic ratio measurements compared amongst the study groups of different leiomyoma localizations (submucous, intramural, subserous) and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided